CLINICAL TRIAL: NCT01004705
Title: Cardiovascular Fixed Dose Combination Pill: A Pharmacodynamic Study of a Fixed Dose Combination of Acetylsalicylic Acid, Simvastatin, and Ramipril in Subjects With Elevated LDL Cholesterol
Brief Title: A Pharmacodynamic Study to Evaluate the Effect of a Fixed Dose Combination Pill on Low Density Lipoprotein (LDL) Cholesterol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P-080647-01
Record Dates: First submitted 2009-10-23; First posted 2009-10-30 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Elevated LDL Cholesterol
Keywords: cardiovascular; fixed; dose; combination; pill; LDL; cholesterol
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Blood Circulation; Aspirin; Simvastatin; Ramipril

ARMS (2):
- Fixed Dose Combination Pill (Experimental): Once daily oral dose of combination of acetylsalicylic acid, simvastatin, and ramipril (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 or 10 mg ramipril)
  Interventions: Drug: Cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin and ramipril),
- Simvastatin (Active Comparator): Once daily oral dose of Simvastatin 40 mg
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin and ramipril), — A once daily oral dose of the cardiovascular fixed dose combination pill ( acetylsalicylic acid, simvastatin, ramipril) for 12 weeks.
  Arms: Fixed Dose Combination Pill
Drug: Simvastatin — A once daily oral dose of simvastatin for 12 weeks.
  Arms: Simvastatin

SUMMARY:
This study evaluates the effect on LDL cholesterol of the 3 drugs given together in the cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin, and ramipril) as compared to the effect on LDL cholesterol of simvastatin given alone. Approximately 76 subjects will be screened, 60 randomized in order about 52 subjects to finish the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age
* Previously untreated LDL cholesterol ≥100 mg/dL and ≤180 mg/dL.
* Provide written informed consent.

Exclusion Criteria:

* Subjects with a medical condition requiring chronic pharmacological treatment
* On direct questioning and physical examination have evidence of any clinically significant chronic disease, including known or suspected human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV) infection.
* On direct questioning and physical examination have a medical history or evidence of abuse of drugs.
* Medical history of gastrointestinal bleeding or gastric or duodenal ulcer.
* Systolic pressure ≥140 mmHg or diastolic pressure >89 mmHg requiring hypotensive medication.
* Presence of secondary dyslipidemia.
* Previous use of cholesterol lowering medication.
* Previous coronary artery bypass graft (CABG).
* Previous percutaneous transluminal coronary angioplasty (PTCA) with a drug-eluting stent.
* Presence of severe congestive heart failure (New York Heart Classification [NYHC] III IV).
* Presence of untreated or uncontrolled thyroid disease.
* Past or current medical history of asthma or aspirin induced asthma
* Previous hypersensitivity to ACE inhibitors (eg angioedema or cough).
* Previous hypersensitivity to ARBs.
* History of unstable angina.
* Serum creatinine >2 mg/dL.
* Creatine phosphokinase (CPK) ≥5 x the upper limit of normal (ULN).
* Hemoglobin ≤12 g/dL (120 g/L) for male subjects or ≤10 g/dL (100 g/L) for female subjects.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 x ULN.
* Total bilirubin ≥1.5 x ULN.
* Serum triglyceride concentration ≥400 mg/dL.
* Subjects not using effective contraception methods (intra uterine device [IUD] and condom or diaphragm with spermicide and condom) during the study and for at least one month thereafter.
* Pregnant, lactating, breastfeeding, or intends to become pregnant during the course of the study (females only). All women must have a negative urine pregnancy test at the Screening Visit, be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or have a postmenopausal status (no menses) for at least one year.
* Contraindications to or known or suspected hypersensitivity to aspirin, simvastatin or ramipril or their excipients.
* Presence of mental illness limiting the capacity for self-care.
* Presence of major systemic illnesses: renal disease, liver disease, neurological or psychiatric disease.
* Participation, in the 30 days preceding enrolment into the study, in any other clinical study in which investigational or marketed drugs were employed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 subjects were screened, 47 met eligibility requirements and 44 entered the run-in period.
Groups:
- Pre-randomization Run-In: Screening period with ramipril 2.5 mg
- Combination Pill Then Simvastatin: After randomization, in Period 1 participants received a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 11 weeks; participants received no intervention during wash-out; in Period 2 participants received a once daily oral dose of 40 mg simvastatin for 12 weeks
- Simvastatin Then Combination Pill: After randomization, in Period 1 participants received a once daily oral dose of 40 mg simvastatin for 12 weeks; participants received no intervention during wash-out; in Period 2 participants received a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 11 weeks.
Period: Run-In
Arm/Group | Pre-randomization Run-In | Combination Pill Then Simvastatin | Simvastatin Then Combination Pill
Started | 44 | 0 | 0
Completed | 36 | 0 | 0
Not Completed | 8 | 0 | 0
Period: Period 1 (12 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Simvastatin | Simvastatin Then Combination Pill
Started | 0 | 18 | 18
Completed | 0 | 13 | 13
Not Completed | 0 | 5 | 5
Period: Washout Period (6 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Simvastatin | Simvastatin Then Combination Pill
Started | 0 | 13 | 13
Completed | 0 | 13 | 13
Not Completed | 0 | 0 | 0
Period: Period 2 (12 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Simvastatin | Simvastatin Then Combination Pill
Started | 0 | 13 | 13
Completed | 0 | 13 | 9
Not Completed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Randomized Patients: All patients randomized to both study sequences (Combination Pill then Simvastatin and Simvastatin then Combination Pill)
Arm/Group | Randomized Patients
Number analyzed (Participants) | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: The Difference in LDL Cholesterol Levels Between the Basal and the Final Visit of Each Treatment Period.
Description: Change from baseline in LDL cholesterol level following each Treatment Period was defined as the difference between the measurements from the baseline visit (Visit 4, Day 1) and Visit 9 (Day 84) for Treatment Period 1, and between the Visit 11 (Day 126) and Visit 16 (Day 210) for Treatment Period 2.
Time Frame: Day 1 and Day 84 of the Period 1 and Day 126 and Day 210 of Period 2
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Combination Pill: Once daily oral dose of combination pill containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril for 11 weeks.
- Simvastatin: Once daily oral dose of 40 mg simvastatin for 12 weeks
Arm/Group | Combination Pill | Simvastatin
Number analyzed (Participants) | 21 | 21
mg/dL | -34.24 (27.103) | -27.95 (32.597)

2. Secondary Outcome: The Difference in Mean Total Cholesterol Between the Basal and the Final Visit of Each Treatment Period.
Description: Change from baseline in mean total cholesterol level following each Treatment Period was defined as the difference between the measurements from the baseline visit (Visit 4, Day 1) and Visit 9 (Day 84) for Treatment Period 1, and between the Visit 11 (Day 126) and Visit 16 (Day 210) for Treatment Period 2.
Time Frame: Day 1 and Day 84 of the Period 1 and Day 126 and Day 210 of Period 2
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Combination Pill | Simvastatin
Number analyzed (Participants) | 21 | 21
mg/dL | -36.81 (28.715) | -29.81 (38.407)

ADVERSE EVENTS:
Time Frame: 36 weeks
Groups:
- Combination Pill: Combination pill containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril for 11 weeks
Arm/Group | Pre-randomization Run-In | Combination Pill | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/44 | 1/31 | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-randomization Run-In (N=44) | Combination Pill (N=31) | Simvastatin (N=31)
Blood phosphokinase creatine increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication must be agreed upon with the sponsor.